CLINICAL TRIAL: NCT04618666
Title: Laparoscopic Versus Open Appendectomy in the Management of Chronic Appendicitis
Brief Title: Laparoscopic Versus Open Appendectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mena helmy, Assistant Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lap appendectomy
Record Dates: First submitted 2020-09-18; First posted 2020-11-06 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-11

CONDITIONS: Chronic Inflammation of Appendix
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: single group in which half of them will be operated open and the other half laparoscopic
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laparoscopic and open appendectomy (Experimental): comparative study between laparoscopic and open appendectomy
  Interventions: Procedure: laparoscopic and open surgery intervention

INTERVENTIONS:
Procedure: laparoscopic and open surgery intervention — laparoscopic and open surgery to remove an inflammed appendix in chronic appendicitis

SUMMARY:
comparison between laparoscopic and open appendectomy in the management of chronic appendicitis

DETAILED DESCRIPTION:
The appendix is a blind-ended tube connected to the cecum, from which it develops in the embryo. The most common diseases of the appendix (in humans) are appendicitis and carcinoid tumors. Appendicitis is inflammation of the appendix. Symptoms commonly include right lower abdominal pain, nausea, vomiting, and decreased appetite. However, approximately 40% of people do not have these typical symptoms . Appendicitis is caused by a blockage of the hollow portion of the appendix. This is most commonly due to a calcified "stone" made of feces. Inflamed lymphoid tissue from a viral infection, parasites, gallstone, or tumors may also cause the blockage. This blockage leads to increased pressures in the appendix, decreased blood flow to the tissues of the appendix, and bacterial growth inside the appendix causing inflammation. The combination of inflammation, reduced blood flow to the appendix and distention of the appendix causes tissue injury and tissue death. If this process is left untreated, the appendix may burst, releasing bacteria into the abdominal cavity, leading to increased complications. The surgical procedure for the removal of the appendix is called an appendicectomy. Appendicectomy can be performed through open or laparoscopic surgery. The surgical procedure for the removal of the appendix is called an appendicectomy . Appendicectomy can be performed through open or laparoscopic surgery. When the surgeon uses the open approach, he makes an incision in the lower right section of the abdomen. Most incisions are less than 3 in (7.6 cm) in length. The surgeon then identifies all of the organs in the abdomen and examines them for other disease or abnormalities. The appendix is located and brought up into the wounds. The surgeon separates the appendix from all the surrounding tissue and its attachment to the cecum, and then removes it. The site where the appendix was previously attached, the cecum, is closed and returned to the abdomen The muscle layers and then the skin are sewn together . When the surgeon performs a laparoscopic appendectomy, four incisions, each about 1 in (2.5 cm) in length, are made. One incision is near the umbilicus, or navel, and one is between the umbilicus and the pubis. Two other incisions are smaller and are on the right side of the lower abdomen. The surgeon then passes a camera and special instruments through these incisions. With the aid of this equipment, the surgeon visually examines the abdominal organs and identifies the appendix. The appendix is then freed from all of its attachments and removed. The place where the appendix was formerly attached, the cecum, is stitched. The appendix is removed through one of the incisions. The instruments are removed and then all of the incisions are closed . The primary objective of this study was to compare the laparoscopic approach and the conventional technique in the treatment of chronic Appendicitis.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of chronic appendicitis - - -Male or Female patients with chronic appendicitis

* Patients who are fit for laparoscopy and general anaeshesia
* Patients who provide a written informed concent
* Patient who agree to provide short term outcome data and agree to provide

Exclusion Criteria - - -Patients with severe comorbid conditions with high risk for general anesthesia.

* Patients suffering from an ongoing infections including chest infections .
* Patients who didn't give concent .
* Children and pregnant women
* Cases of complicated appendicitis .

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
assesment of operative time | 1 hour
  discover whether open or laparoscopic appendectomy takes longer time